CLINICAL TRIAL: NCT00043316
Title: A Phase I/II Study of Interferon Gamma-1b by Inhalation for the Treatment of Patients With Cystic Fibrosis
Brief Title: Interferon Gamma-1b by Inhalation for the Treatment of Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: InterMune (Industry)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GICF-001
Record Dates: First submitted 2002-08-07; First posted 2002-08-09 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; pulmonary impairment
MeSH Terms: conditions — Cystic Fibrosis | interventions — interferon gamma-1b

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: interferon gamma-1b — 500 or 1000 mcg, inhalation, 3x per week

SUMMARY:
The purpose of this research study is to evaluate the safety and effectiveness of Interferon gamma-1b (IFN-g 1b) on lung function when given to patients with cystic fibrosis by inhalation (breathed into the lungs) three times a week for 12 weeks.

The FDA has not approved Interferon gamma-1b for use with cystic fibrosis patients, which is the condition being examined in this study.

ELIGIBILITY:
Key inclusion criteria:

* At least 12 years of age
* Diagnosis of cystic fibrosis with mild to moderate pulmonary impairment
* Must be receiving ongoing chronic treatment with TOBI (inhaled tobramycin) OR not receiving ongoing chronic treatment with TOBI and no use of TOBI or other inhaled antibiotic within 4 weeks prior to study drug administration·
* Other specific diagnostic indicators of CF and other factors must meet minimum requirements.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2001-02; Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
change in FEV1, sputum bacterial density | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steve Porter, MD, Study Director — InterMune
Locations (17):
- United States (17):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Palo Alto, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Denver, Colorado
  - Daytona Beach, Florida
  - Orlando, Florida
  - Chicago, Illinois
  - New Orleans, Louisiana
  - Rochester, Minnesota
  - New York, New York
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Lackland Air Force Base, Texas
  - Tyler, Texas